CLINICAL TRIAL: NCT00944658
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Apremilast (CC-10004)in the Treatment of Ankylosing Spondylitis (AS)
Brief Title: Spondylitis Trial of Apremilast for Better Rheumatic Therapy
Acronym: START
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112008; 2008-004229-40 (EudraCT Number)
Record Dates: First submitted 2009-07-20; First posted 2009-07-23 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; Imaging
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — apremilast; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo twice a day for 12 weeks, 4 weeks follow up
  Interventions: Drug: Placebo (sugar pill)
- Apremilast (Active Comparator): 30 mg twice a day for 12 weeks, 4 weeks follow up
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 10mg twice a day, dose was titrated by 20mg every 2 days until the maximum dose 30mg twice a day for 12weeks
  Arms: Apremilast
Drug: Placebo (sugar pill) — twice a day
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of apremilast in AS as measured by improvement in patients' signs and symptoms of the disease and changes in imaging. Additionally the safety and tolerability of apremilast in AS will be assessed.

DETAILED DESCRIPTION:
Presently, there are very few treatments available which affect the progression of the disease in the spine. The only proven treatment is the use of drugs inhibiting tumour necrosis factor alpha (TNF). However, there are limitations with this treatment in that it needs to be administered via an injection and is also very expensive. Therefore it is necessary to develop new therapeutic agents for this condition.

Apremilast (the study drug) is an oral tablet which has been shown to inhibit TNF production in a mouse model of inflammation. It has also been used in clinical trials for asthma and psoriasis in humans with good affect and tolerability.

These studies were funded by Celgene Corporation and they will be funding this study.

The patients will be recruited from hospitals by Consultant referral. The patients will have had AS for at least 2 years and their symptoms will have been uncontrolled on conventional non-steroidal anti-inflammatory drugs such as ibuprofen. Patients will be randomised to either receive apremilast or a placebo and treated over a period of 12 weeks. They will then be followed up for 28 days after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this trial
* Diagnosis of ankylosing spondylitis as defined by the modified New York criteria (1984) as follows:

  1. a history of inflammatory back pain;
  2. limitation of motion of the lumbar spine in both the sagittal and frontal planes;
  3. limited chest expansion, relative to standard values for age and sex;
  4. definite radiographic / imaging evidence of sacroiliitis and/or spinal inflammation
* Patients must have daily spinal pain and stiffness for at least 2 weeks prior to randomization. This is defined by having a score of >1 on questions #2 and #5 of the BASDAI score for the 2 weeks prior to randomization.
* Patients receiving NSAIDS and/or COX-2 inhibitors must be on stable doses for at least 2 weeks prior to randomization.
* Age >18 years
* Male and female patients, who are not surgically sterile or postmenopausal, must use reliable methods of birth control for the duration of the study. Males must agree to use barrier contraception for 3 months following the end of the trial.
* Women of childbearing potential, not surgically sterile or postmenopausal, must have a negative serum beta HCG.

Exclusion Criteria:

* Use of DMARDs (methotrexate, d-penicillamine, sulfasalazine, azathioprine, hydroxychloroquine, or gold) within 8 weeks of randomization.
* Use of systemic corticosteroids within 4 weeks of randomization
* Use of intravenous or intra-articular corticosteroids within 4 weeks of randomization
* Use of TNF alpha blockers (eg, infliximab, adalimumab) or etanercept as follows:

Compound PK Exclusion period Etanercept T ½ = 102 hrs = 4.25 days 4 weeks Adalimumab T ½ 2 wks; 5 half lives 10 weeks 10 weeks Infliximab T ½ 7.7-9.5 d 12 weeks 8 weeks after maintenance dose median infx conc 0.5-6 mcg/ml

* Therapy with an investigational agent within 30 days of randomization or 5 half-lives (pharmacokinetic or pharmacodynamic), which ever is longer
* Known HIV or hepatitis B or C infection
* Exclusion of tuberculosis (TB)

  * History of active Mycobacterium tuberculosis infection (any subspecies) within 3 years prior to the screening visit. Infections that occurred > 3 years prior to entry must have been effectively treated.
  * History of incompletely treated latent Mycobacterium tuberculosis infection (as indicated by a positive Purified Protein Derivative [PPD] skin test)
  * Clinically significant abnormality on chest x-ray (CXR) if mantoux >5mm or ELISPOT positive
* History of other rheumatic autoimmune diseases (eg, systemic lupus erythematosus, rheumatoid arthritis, etc.)
* Pregnant or nursing women
* Any condition, in the investigator's opinion, which places the patient at an undue risk by participating in the study.
* Contraindication to MRI and other MRI exclusions following local centre guidelines (Appendix H)
* An estimated glomerular filtration rate (eGFR) of < 60 ml/min (because of the small risk of nephrogenic sclerosing fibrosis with gadolinium intravenous contrast), if patient is to have MRI with gadolinium contrast .
* Claustrophobia
* Hemoglobin < 9 g/dL
* White blood cell (WBC) count < 3000 /μL (≥ 3.0 X 109/L) and ≥ 14,000/μL (≥ 20 X 109/L)
* Neutrophils < 1500 /μL (< 1.5 X 109/L)
* Platelets < 100,000 /μL (< 100 X 109/L)
* Serum creatinine > 1.5 mg/dL (> 132.6 μmol/L)
* Total bilirubin > 2.0 mg/dL
* Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) > 1.5x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Taylor, Principal Investigator — Imperial College London
Locations (1):
- The Kennedy Institute Clinical Trials Unit, 4 West, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pathan E, Abraham S, Van Rossen E, Withrington R, Keat A, Charles PJ, Paterson E, Chowdhury M, McClinton C, Taylor PC. Efficacy and safety of apremilast, an oral phosphodiesterase 4 inhibitor, in ankylosing spondylitis. Ann Rheum Dis. 2013 Sep 1;72(9):1475-80. doi: 10.1136/annrheumdis-2012-201915. Epub 2012 Sep 14. PMID 22984171

RESULTS

PARTICIPANT FLOW:
Period: Treatment 12 Weeks
Arm/Group | Placebo | Apremilast
Started | 19 | 19
Completed | 19 | 17
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Follow up 4 Weeks
Arm/Group | Placebo | Apremilast
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.21 (13.3) | 44.88 (11.1) | 42.95 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 17 | 15 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19 | 17 | 36
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) [Mean (Standard Deviation); unit: units on a scale] — The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue, 0 being no problem and 10 being the worst problem
  units on a scale | 4.36 (1.75) | 4.79 (2.16) | 4.57 (1.95)
Bath Ankylosing Spondylitis Functional Index (BASFI) [Mean (Standard Deviation); unit: units on a scale] — A visual analogue scale with 0 being "easy" and 10 "impossible"
  units on a scale | 3.19 (2.2) | 4.55 (2.42) | 3.87 (2.31)
CRP C-reactive protein [Mean (Standard Deviation); unit: mg/dl] | 6.24 (2.56) | 11.37 (12.12) | 8.8 (7.34)

OUTCOME MEASURES:

1. Primary Outcome: Changes of Apremilast in Patients With AS, Changes in BASDAI Score From Baseline
Description: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), 0 - 10 score, higher reduction in the scores suggest better suboptimal control of disease.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 19 | 17
units on a scale | -0.77 (1.47) | -1.59 (1.48)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p = 0.139, ANCOVA

2. Primary Outcome: Changes of Apremilast on the Signs and Symptoms of AS, Night Pain From Baseline
Description: This endpoint the night time pain score change was recorded by questionnaire to evaluate the Apremilast effect on symptom, higher reduction better improvement.
  scale is 0-10
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 19 | 17
score on a scale | -0.23 (2.75) | -0.81 (3.01)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p = 0.58, ANCOVA

3. Primary Outcome: Effect of Apremilast in Patients With AS, Changes in BASFI Score
Description: Bath Ankylosing Spondylitis Functional Index (BASFI), 0 - 10 score, higher reduction in the scores suggest better suboptimal control of disease.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 19 | 17
units on a scale | -0.28 (1.61) | -1.74 (1.91)
Statistical Analysis 1: Comparison: Placebo vs Apremilast; Test type: Superiority; p = 0.108, ANCOVA; Rank Ancova

4. Secondary Outcome: The Safety and Tolerability of Apremilast in AS, Number of Participants With Adverse Events
Description: To evaluate the safety and tolerability of Apremilast in AS, the investigator recorded the incidence of adverse events.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 19 | 19
Participants | 17 | 18

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Placebo | Apremilast
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 17/19 | 18/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Apremilast (N=19)
Headache (Nervous system disorders) | 5 (5) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 6 (6)
Loose stools (Gastrointestinal disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Flatulance (Gastrointestinal disorders) | 0 (0) | 2 (2)
raised serum amylase (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Diarrhoe (Gastrointestinal disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
It was most likely underpowered to detect a signiﬁcant beneﬁt of Apremilast in AS patients because no information on an effect size was available to aid in the study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes